CLINICAL TRIAL: NCT03991988
Title: Effects of Montelukast Therapy on Alzheimer's Disease (EMERALD)
Brief Title: Montelukast Therapy on Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ihab Hajjar, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00111553
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer
MeSH Terms: conditions — Alzheimer Disease | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montelukast Group (Experimental): Montelukast (10, 20, or 40 mg)
  Interventions: Drug: Montelukast
- Placebo Group (Placebo Comparator): Matched placebo pill
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Montelukast — Participants in this arm will take a pill of Montelukast daily on escalating doses: 10, 20 to 40 mg.
  All participants will be initiated on 10 mg. The dose will be increased in 2-week increments to 20 mg and 40 mg as long as participants report no intolerable symptoms or adverse events.
  Arms: Montelukast Group
Drug: Placebo oral tablet — Participants in this arm will take a matched placebo pill daily
  Arms: Placebo Group

SUMMARY:
This is a one-year, double-blind placebo-controlled randomized clinical trial that compares montelukast to placebo in individuals with mild cognitive impairment (MCI) and early Alzheimer's disease (AD) dementia. The measures include cognitive function, cerebrospinal fluid (CSF) biomarkers and neuroimaging (cerebral perfusion and markers of vascular brain damage).

Participants will be treated with montelukast (escalating doses:10, 20 to 40 mg) or matched placebo.

DETAILED DESCRIPTION:
Treatment options for Alzheimer's disease (AD) remain limited, especially treatments linking neurovascular and neuroinflammatory changes with clinical manifestations of the disease. Prior research studies have documented a positive effect of cysteinyl leukotriene type 1 (cysLT-1) receptor antagonist, particularly Montelukast, on inflammatory processes in the brain and on neuronal injury, blood-brain-barrier (BBB) integrity, and amyloid-β42 (Aβ) protein accumulation. Although montelukast is currently in use for the treatment of inflammatory diseases e.g. bronchial asthma and exercise-induced bronchospasm, its effects on memory and thinking abilities and on AD biomarkers are yet to be fully understood.

This is a single site randomized controlled trial at Emory University that compares the effects of montelukast vs. placebo on memory and thinking abilities, as well as on brain imaging and markers of brain degeneration. Each participant will undergo a screening process following informed consent to determine if they meet study eligibility criteria. Participants will be enrolled in the study for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 50 years or older
2. MCI group will be defined based on:

   (i) Subjective memory concern;

   (ii) Abnormal memory function documented using the Logical Memory subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale-Revised (the maximum score is 25): [<11 for 16 or more years of education; <9 for 8-15 years of education; <6 for <7 years of education];

   (iii) Montreal Cognitive Assessment (MoCA) < 26;

   (iv) Clinical Dementia Rating (CDR) scale /Memory box score=0.5;

   (v) General functional performance sufficiently preserved (Functional Assessment Questionnaire ≤5).
3. Early AD dementia group will be defined based on:

   (i) Subjective memory concern;

(ii) Abnormal memory function documented using the Logical Memory subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale-Revised (the maximum score is 25): [<11 for 16 or more years of education; <9 for 8-15 years of education; <6 for <7 years of education];

(iii) Montreal Cognitive Assessment (MoCA) <26;

(iv) Clinical Dementia Rating scale/Memory box score 1 or 2;

(v) Early AD dementia defined as Functional Assessment Staging Test (FAST) of 4 or 5

Exclusion Criteria:

1. Intolerance to Montelukast;
2. Current diagnosis of bronchial asthma or exercise-induced bronchospasm and currently on Montelukast or other leukotriene receptor antagonists (Zafirlukast, Pranlukast);
3. Liver disease (elevated liver enzymes (>2x normal): Alanine aminotransferase (ALT), AST, alkaline phosphatase, total bilirubin);
4. Renal disease (Creatinine >2.0 mg/dl), platelets<50,000/μl, or INR>1.9;
5. Diagnosis of any neurological or psychiatric disorders that affects cognition such as uncontrolled depression, schizophrenia, Parkinson's disease or use of anti-Parkinsonian therapies (unless used for essential tremor), multiple sclerosis, or other active medical condition that in the judgment of the study physicians would affect the safety of the subject or scientific integrity of the study;
6. Other contributing factors to cognitive impairment such as uncontrolled hypothyroidism (TSH >10 mU/l) or untreated low vitamin B12 (<250 ng/mL);
7. Uncontrolled congestive heart failure reflected by poor exercise tolerance and shortness of breath at rest or with some exertion;
8. Actively undergoing chemotherapy or radiation therapy for cancer treatment;
9. History of stroke in the past 3 years;
10. Severely impaired cognition (MoCA ≤10, FAST >5 or CDR >2);
11. Inability to have MRI and LP e.g. for MRI, metal implants or cardiac pacemaker or for LP, bleeding diathesis from disease states or from use of anticoagulants such as warfarin, heparin and related products, Rivaroxaban or Xarelto, Apixaban or Eliquis, Edoxaban or Savaysa, Dabigatran or Pradaxa. Subjects who can have either one lumbar puncture (LP) or MRI will be enrolled;
12. Inability to have cognitive assessment due to hearing, vision, or language issues or due to severe impairment;
13. History of increased intracranial pressure (ICP);
14. In those who are unable to demonstrate that they understood the details of the study using the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) instrument modified for EMERALD (i.e. lack of decisional-capacity to consent), a study partner/surrogate who can sign on their behalf will be required; otherwise, they will be excluded;
15. Use of phenobarbital or rifampin due to drug interaction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Hajjar, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital Clinical Research Network, Atlanta, Georgia
  - Executive Park, Atlanta, Georgia
  - Wesley Woods, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast Group: Montelukast (10, 20, or 40 mg)
  Montelukast: Participants in this arm will take a pill of Montelukast daily on escalating doses: 10, 20 to 40 mg.
  All participants will be initiated on 10 mg. The dose will be increased in 2-week increments to 20 mg and 40 mg as long as participants report no intolerable symptoms or adverse events.
Period: Overall Study
Arm/Group | Montelukast Group | Placebo Group
Started | 16 | 16
Completed | 14 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast Group | Placebo Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.8) | 73.9 (7.7) | 72.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 12 | 16 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Mild Cognitive Impairment (MCI) [Count of Participants; unit: Participants] | 10 | 9 | 19
Dementia [Count of Participants; unit: Participants] | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Gastrointestinal (GI) Symptoms
Description: Number of participants with any GI symptoms reported: diarrhea, nausea, vomiting
Time Frame: Baseline, 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 16
Participants | 1 | 1

2. Primary Outcome: Number of Participants With Reported Anaphylaxis
Description: Number of participants with reported anaphylaxis during follow up time
Time Frame: Baseline, 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 16
Participants | 1 | 0

3. Primary Outcome: Number of Participants With Elevated Liver Enzymes
Description: Number of participants with elevated liver enzymes during follow up
Time Frame: Baseline, 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

4. Primary Outcome: Prothrombin Time (PT)/ International Normalized Ratio (INR)
Description: Prothrombin time (PT)/ international normalized ratio (INR) will be measured at baseline and 1 year.
Time Frame: Baseline, 1 year
Population: Data captured from participants with CSF data or who completed a lumbar puncture procedure and have available results for PT/INR.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 11 | 12
ratio
  Baseline: number analyzed (Participants) | 11 | 10
  Baseline | 1.05 (0.02) | 1.02 (0.01)
  1 year: number analyzed (Participants) | 0 | 2
  1 year |  | 1.05 (0.05)

5. Primary Outcome: Neuropsychiatric Inventory Questionnaire (NPI-Q) Score
Description: The NPI-Q is designed to be a self-administered questionnaire completed by informants about patients for whom they care. Each of the 12 NPI-Q domains contains a survey question that reflects cardinal symptoms of that domain. Initial responses to each domain question are "Yes" (present) or "No" (absent). If the response to the domain question is "No", the informant goes to the next question. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale and the associated impact of the symptom manifestations on them (i.e. Caregiver Distress) using a 5-point scale. The NPI-Q provides symptom Severity and Distress ratings for each symptom reported, and total Severity and Distress scores reflecting the sum of individual domain scores. NPI-Q Severity score range: 0-36 (lower is better).
Time Frame: Baseline, 1 year
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline | 5.00 (0.97) | 2.62 (0.95)
  1 year | 5.68 (1.04) | 2.73 (1.02)

6. Primary Outcome: Number of Patients With Seizures
Description: Number of participants that reported seizures during follow up time
Time Frame: Baseline, 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

7. Primary Outcome: Number of Discontinuations From Montelukast
Description: Number of participants that stopped taking Montelukast during follow up time
Time Frame: Baseline, 1 year
Population: This outcome measured the number of participants that stopped taking Montelukast. This outcome was not assessed in the Placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 0
Participants | 0 | 0

8. Secondary Outcome: CSF Amyloid
Description: A lumbar puncture will be done at baseline and at 12 months follow up Approximately 30-45 ml of CSF will be collected using sterile polypropylene collection tubes.
  Amyloid-β42 is reported as pg/ml.
Time Frame: Baseline, 1 year
Population: 22 participants with CSF amyloid data captured (11 in Montelukast group and 11 in placebo group).
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 11 | 11
pg/ml
  Baseline | 849.4 (77.34) | 704.6 (89.48)
  1 year | 795.5 (76.60) | 695.2 (88.11)

9. Secondary Outcome: CSF Tau Levels
Description: CSF tau protein (CSF-tau) is found in most patients with Alzheimer's disease. A lumbar puncture will be done at baseline and at 12 months follow up. Approximately 30-45 ml of CSF will be collected using sterile polypropylene collection tubes. Results will be reported as Phospho tau (p-tau181) in pg/ml.
Time Frame: Baseline, 1 year
Population: 22 participants with CSF tau data captured (11 in Montelukast group and 11 in placebo group).
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 11 | 11
pg/ml
  Baseline | 20.6 (2.42) | 22.8 (2.81)
  1 year | 21.1 (2.48) | 21.9 (2.86)

10. Secondary Outcome: Clinical Dementia Rating (CDR) Score
Description: The CDR rates each of the six general domains (or boxes) involving memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care, and a global rating is then generated, ranging from 0 to 3. A score of 0 = normal, 0.5 = very mild dementia, 1 = mild dementia, 2 = moderate dementia, and 3 = severe dementia.
Time Frame: Baseline, 1 year
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline | 0.6 (0.05) | 0.6 (0.04)
  1 year | 0.7 (0.07) | 0.7 (0.07)

11. Secondary Outcome: NIH Toolbox Cognition Battery (NIHTB-CB)
Description: The NIH Toolbox® is a computer-based comprehensive set of neuro-behavioral measurements that reliably and validly assesses neurocognitive sub-domains in clinical trials, including working memory, episodic memory, processing speed, language, attention and executive function. The fluid cognitive composite (FCC) score is derived by averaging the standard scores of each of the fluid tests (Picture Sequence Memory, List Sorting, Pattern Comparison, Flanker, and Dimensional Change Card Sort.), and then deriving standard scores based on this new distribution. The fully-adjusted FCC T-score is reported. Higher score indicates with better performance. The score ranged from a minimum of 19 (0th percentile) to a maximum of 58 (79th percentile) in this sample. The population-level T-score and percentile rank range from 23 (0.3th percentile) to 77 (99.6th percentile) with mean=50 and SD=10.
Time Frame: Baseline, 1 year
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Montelukast Group | Placebo Group
Number analyzed (Participants) | 16 | 16
t-score
  Baseline | 35.2 (2.53) | 35.4 (2.93)
  1 year | 33.9 (2.89) | 37.3 (3.41)

ADVERSE EVENTS:
Time Frame: During follow up time, an average of 1 year
Description: All participants on the Montelukast arm with reported AEs were safely escalated to 40 mg dose, and all their AEs resolved spontaneously with no sequelae. AE results were collected altogether (not dose based).
Groups:
- Montelukast Group: Montelukast (10, 20, or 40 mg)
  Montelukast: Participants in this arm will take a pill of Montelukast daily on escalating doses: 10, 20 to 40 mg.
  All participants were initiated on 10 mg, and the dose increased in 2-week increments to 20 mg and 40 mg as long as participants report no intolerable symptoms or adverse events.
Arm/Group | Montelukast Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast Group (N=16) | Placebo Group (N=16)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Low Mood (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A limitation of the study is its relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT03991988/Prot_SAP_000.pdf